CLINICAL TRIAL: NCT06526520
Title: Relaxin Measurement in Different Endometrial Preparation Approaches for Frozen Embryo Transfer
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2406-ABU-007-BL
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Frozen Embryo Transfer
Keywords: frozen embryo transfer; hormonal replacement cycle; natural cycle; Relaxin

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests for hormonal assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Natural cycle: Monitoring of a natural cycle
- natural proliferative phase cycle: Monitoring of a natural proliferative phase cycle
  Interventions: Drug: Exposure to progesterone or HRT medication
- Hormonal replacement cycle: Monitoring of a hormonal replacement cycle
  Interventions: Drug: Exposure to progesterone or HRT medication

INTERVENTIONS:
Drug: Exposure to progesterone or HRT medication — to add either progesterone only in the NPP protocol or E2 and progesterone in a HRT protocol
  Groups: Hormonal replacement cycle; natural proliferative phase cycle

SUMMARY:
To investigate the levels of Relaxin in different types of endometrial preparation for a frozen embryo transfer cycle. Up to now it is unclear, whether ovulation with a functional corpus luteum (CL) will be present in a natural proliferative phase (NPP) endometrial preparation approach.

DETAILED DESCRIPTION:
The last years have seen a distinct shift from fresh (fresh ET) to frozen embryo transfer (FET) cycles. Furthermore it became obvious, that the endometrial preparation approach has a significant impact on the course of the pregnancy and that a HRT endometrial preparation approach is associated with a higher risk for bleeding and miscarriages in early pregnancy and for the development of pregnancy induced hypertension and pre-eclampsia later in pregnancy.

These conditions are attributed to the absence of a CL in the HRT approach. Lately a new endometrial preparation approach is discussed and performed, the so called natural proliferative phase protocol, in which the follicle growth is monitored and when the lining is deemed to have a sufficient thickness and the triple lining pattern, exogeneous progesterone is started to induce secretory transformation before spontaneous ovulation. Despite some studies showing, that exogeneous progesterone administration might induce ovulation, it is not clear whether there will be a CL, producing Relaxin, in the NPP approach.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles

Exclusion Criteria:

* abnormal findings of the ovaries (e.g endometriosis)
* Intake of any hormones within 3 months of study start
* desire to become pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — regular menstrual cycles
Study Population: - healthy volunteers with regular cycles
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relaxin measurement | 4 to 6 months
  Measurement of Relaxin in the different types of frozen embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — ART Fertility Clinic
Locations (1):
- ART Fertiltiy Clinic, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
on request